CLINICAL TRIAL: NCT05853445
Title: A Prospective, Non-interventional Study of JAKAVI® (Ruxolitinib) Treatment in Patients With Polycythemia Vera (PAVE)
Brief Title: A Prospective, Non-interventional Study of JAKAVI® (Ruxolitinib) Treatment in Patients With Polycythemia Vera
Acronym: PAVE
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC424BDE12
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Polycythemia Vera
Keywords: ruxolitinib; polycythemia vera; PV; jakavi
MeSH Terms: conditions — Polycythemia Vera | interventions — ruxolitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- JAK inhibitor naive: JAK inhibitor naive patients
  Interventions: Other: Jakavi
- JAK inhibitor pre-treated: JAK inhibitor pre-treated patients (Jakavi® or any other JAK inhibitor for ≥3 months)
  Interventions: Other: Jakavi

INTERVENTIONS:
Other: Jakavi — Prospective observational study. There is no treatment allocation. Patients administered Jakavi by prescription and administered according to the SmPC.
  Other Names: Ruxolitinib

SUMMARY:
Jakavi® therapy for polycythemia vera (PV) has so far been studied exclusively in clinical trials and at selected clinical trial centres. This observational study is intended to document the therapy of PV in daily practice with a broad patient population and a geographically representative selection of German centres (both hospitals and practices). The prospective mapping of daily practice reality is thus the main goal of this project.

DETAILED DESCRIPTION:
To achieve meaningful results in accordance with the study objective and to obtain long-term data from daily clinical practice in a real-world setting, the observation period under Jakavi® therapy is specified as 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients with PV for whom Jakavi® therapy is indicated according to the European summary of product characteristics
* Patients who have been informed about this NIS and gave written consent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients with PV for whom Jakavi® therapy is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Dosing | Up to 36 months
  Number of patients by initial dosing and number of patients with dose modifications will be provided
Treatment interruptions | Up to 36 months
  Number of patients with treatment interruptions
Overall survival | Up to 36 months
  Overall survival for JAK inhibitor naive and pretreated patients
Hematology | Up to 36 months
  Number of patients with changes in different blood count values over time (hematocrit, erythrocytes, thrombocytes, leukocytes)
Number of phlebotomies | Up to 36 months
  Total number of phlebotomies
Change in spleen size (or volume) | Up to 36 months
  Measured by palpation/sonography/CT/MRI
Quality of Life (QoL) - MPN-SAF TSS; MPN-10 | Up to 36 months
  The Myeloproliferative Neoplasm (MPN) Symptom Assessment Form Total Symptom Score (MPN-SAF TSS; MPN-10) questionnaire contains the ten most clinically relevant symptoms reported by patients with MPNs.
  It includes disease related symptoms each scored from 0 (absent) to 10 (worst imaginable). Total Scores range from 0-100, with higher scores indicating a greater number of symptoms and severity.
Thromboembolic events | Up to 36 months
  Number of patients with thromboembolic events.

SECONDARY OUTCOMES:
Eastern Cooperative Oncology Group (ECOG) performance status | Up to 36 months
  The ECOG performance status is a scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  The grade ranges from 0 (fully active, able to carry on all pre-disease performance without restriction) to 5 (dead)
Change in constitutional symptoms | Up to 36 months
  Number of patients with change in constitutional symptoms
Quality of Life (QoL) - (SF-36) | Up to 36 months
  The Short Form-36 questionnaire consists of questions measuring physical function, physical role limitation, pain, general health, vitality, social function, emotional role limitations, and mental health status. The scores that can be obtained from the scale vary between 0 and 100 and the increase in the scores indicates that the quality of life is high.
Bone marrow aspiration and biopsy | Up to 36 months
  Number of Biopsies per visit
Molecular examination | Up to 36 months
  Number of performed assessments of JAK2V617F mutation per visist

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (87):
- Germany (87):
  - Novartis Investigative Site, Heidenheim, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Reutlingen, Baden-Wurttemberg
  - Novartis Investigative Site, Winnenden, Baden-Wurttemberg
  - Novartis Investigative Site, Aschaffenburg, Bavaria
  - Novartis Investigative Site, Augsburg, Bavaria
  - Novartis Investigative Site, Donauwörth, Bavaria
  - Novartis Investigative Site, Erlangen, Bavaria
  - Novartis Investigative Site, Herrsching am Ammersee, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Frankfurt (Oder), Brandenburg
  - Novartis Investigative Site, Landshut, Bvaria
  - Novartis Investigative Site, Brake, Lower Saxony
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Twistringen, Lower Saxony
  - Novartis Investigative Site, Duisburg, North Rhine-Westphalia
  - Novartis Investigative Site, Bad Salzuflen, Northrhine Westfalia
  - Novartis Investigative Site, Iserlohn, Northrhine Westfalia
  - Novartis Investigative Site, Bautzen, Saxony
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Pirna, Saxony
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Erfurt, Thuringia
  - Novartis Investigative Site, Altötting
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Soden
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düren
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Fürth
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Halberstadt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hamelin
  - Novartis Investigative Site, Hamm
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Hof
  - Novartis Investigative Site, Idar-Oberstein
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Koblenz
  - Novartis Investigative Site, Kronach
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lemgo
  - Novartis Investigative Site, Loerrach
  - Novartis Investigative Site, Lüdenscheid
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Mayen
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Moers
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Naunhof
  - Novartis Investigative Site, Nordhorn
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Offenburg
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Passau
  - Novartis Investigative Site, Porta Westfalica
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rüsselsheim am Main
  - Novartis Investigative Site, Schorndorf
  - Novartis Investigative Site, Schöneck
  - Novartis Investigative Site, Stolberg
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Westerstede
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Wittenberg
  - Novartis Investigative Site, Wolfsburg
  - Novartis Investigative Site, Würselen
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CINC424BDE12 that is getting linked from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18164